CLINICAL TRIAL: NCT03241004
Title: Does Melatonin Affect Anesthetic MAC (Minimum Alveolar Concentration)?
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: change in study staffing
Sponsor: Englewood Hospital and Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: E-17-705
Record Dates: First submitted 2017-08-02; First posted 2017-08-07 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Anesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive Care Unit (Experimental): Patients will be induced in a standard fashion using intravenous (IV) anesthetics. A continuous administration of propofol will be used for maintenance of anesthesia.
  Baseline EEG readings will be established for 30 minutes, then EEG data will be recorded and a sleep mask applied to the patient for one hour. After one hour, eye masks will be removed for an hour and reapplied after another hour. During the hour that the mask is off, 2 hours into sedation, EEG data will again be recorded.
  Interventions: Other: Sleep Mask
- Operating Room (Experimental): Patients will be induced in a standard fashion using intravenous (IV) anesthetics. A continuous administration of propofol and inhalational anesthetics will be used for maintenance of anesthesia.
  Baseline EEG readings will be established for 30 minutes, then EEG data will be recorded and a sleep mask applied to the patient for one hour. After one hour, eye masks will be removed for an hour and reapplied after another hour. During the hour that the mask is off, 2 hours into sedation, EEG data will again be recorded.
  Interventions: Other: Sleep Mask

INTERVENTIONS:
Other: Sleep Mask — sleep mask applied for two separate 60-minute periods during anesthesia

SUMMARY:
This study aims to determine if anesthetic depth can be deepened non-pharmacologically through use of sleep masks. This study seeks to demonstrate a relationship between the depth of anesthesia with application of sleep masks intraoperatively and in the critical care setting.

DETAILED DESCRIPTION:
Depth of anesthesia will be monitored, both with a standard sleep mask applied and without, in each subject using standard electroencephalogram (EEG) readings via forehead leads and Masimo Sedline 2.0 4-lead EEG monitors.

OR Subjects:

Patients will be induced in a standard fashion using intravenous (IV) anesthetics. A continuous administration of propofol and inhalational anesthetics will be used for maintenance of anesthesia. The standard electroencephalogram (EEG) reading via forehead leads and Masimo Sedline 2.0 4-lead EEG machines will be used to monitor the depth of anesthesia, both with and without the sleep mask.

ICU Subjects:

Patients will be induced in a standard fashion using intravenous (IV) anesthetics. A continuous administration of propofol will be used for maintenance of anesthesia. The standard electroencephalogram (EEG) reading via Masimo Sedline 2.0 4-lead EEG monitors will be used to track the depth of anesthesia, both with and without the sleep mask.

All Subjects:

In both settings,once baseline EEG readings are established (30 minutes), EEG data will be recorded and a sleep mask will be applied to the patient for one hour. After one hour (90 minutes), EEG data will be recorded and the sleep mask will be removed. After another hour (150 minutes), EEG data will be recorded and the mask reapplied. After another hour (210 minutes), EEG data will be recorded and the mask removed. The levels/doses of anesthetic agent at each time point will also be recorded.

Subjective perception of depth of anesthesia will be obtained by means of a post-procedure evaluation administered to each subject.

ELIGIBILITY:
Inclusion Criteria:

* Male or female at least 18 years of age.
* Not pregnant.

Exclusion Criteria:

* Undergoing surgeries expected to last less than 3 hours.
* Undergoing vascular or neurosurgical procedures.
* Patients with history of CVA (Cardiovascular accidents or disease) or other neurological dysfunction.
* Patients or authorized representatives unable or unwilling to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-07-07 (Actual); Primary Completion 2021-07-08 (Actual); Study Completion 2021-07-08 (Actual)

PRIMARY OUTCOMES:
EEG data | 2 hours
  change in depth of anesthesia from baseline to two hours

SECONDARY OUTCOMES:
Subject perception of depth of anesthesia | within 24 hours of reversal of sedation
  post-procedure evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Smok, MD, Principal Investigator — Englewood Hospital and Medical Center
Locations (1):
- Englewood Hospital and Medical Center, Englewood, New Jersey, United States

REFERENCES:
- See also: Related Info — http://www.englewoodhealth.org/for-healthcare-professionals/clinical-research-center